CLINICAL TRIAL: NCT02550977
Title: Multicenter, Open-label, Uncontrolled Study to Investigate Suppression of Ovarian Activity of a Transdermal Contraceptive Patch Containing 0.55 mg Ethinyl Estradiol and 2.1 mg Gestodene in 80 Young Female Volunteers Over 3 Treatment Cycles
Brief Title: Russia/Ukraine Suppression of Ovarian Activity Study
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 16119
Record Dates: First submitted 2015-09-02; First posted 2015-09-16 (Estimated); Last update posted 2017-08-07 (Actual); Status verified 2017-07

CONDITIONS: Contraception
Keywords: Contraception; Transdermal contraceptive patch; Safety; Efficacy; Pharmacokinetic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Gestodene/EE Patch (Experimental)
  Interventions: Drug: Gestodene/EE Patch (BAY86-5016)

INTERVENTIONS:
Drug: Gestodene/EE Patch (BAY86-5016) — 7 day patch containing 0.55 mg ethinyl estradiol and 2.1 gestodene in a 21 day regimen.

SUMMARY:
The purpose of this study is to look into the effectiveness of a new investigational medication applied as a transdermal patch. The patch is applied on the skin with study medication that is absorbed through the skin suppressing ovarian activity and therefore preventing an egg from leaving an ovary (ovulation). The study will look into the study drug's safety and how well it is tolerated and its absorption, breakdown and elimination in the body. It describes how the body affects a specific drug after administration.

ELIGIBILITY:
Inclusion Criteria:

* Healthy female subjects requesting contraception
* Aged 18 to 35 years (inclusive); smokers must not be older than 30 years
* Normal or clinically insignificant cervical smear not requiring further follow-up
* History of regular cyclic menstrual periods
* Willingness to use nonhormonal methods of contraception during the entire study
* Proven ovulation upon completion of the pretreatment cycle

Exclusion Criteria:

* Pregnancy or lactation
* Obesity (body mass index [BMI] > 30.0 kg/m2)
* Significant skin reaction to transdermal preparations or sensitivity to surgical/medical tape
* Any disease or condition that may worsen under hormonal treatment
* Use of hormonal contraception other than study medication during the study

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 91 (Actual)
Dates: Start 2015-09-18 (Actual); Primary Completion 2016-07-15 (Actual); Study Completion 2016-08-15 (Actual)

PRIMARY OUTCOMES:
Suppression of ovulatory activity proved by progesterone and estradiol concentrations | Treatment day 29 to day 84
  Estradiol levels > 100pmol/L indicate some ovarian activity and progesterone levels > 5nmol/L in subjects with estradiol levels > 100pmol/L reflect ovulation or luteinized unruptured follicles.

SECONDARY OUTCOMES:
Serum concentration, AUC (area under curve) of Gestodene | Multiple time points up to treatment day 84
Serum concentration, AUC (area under curve) of ethinyl estradiol | Multiple time points up to treatment day 84
Serum concentration, AUC (area under curve) of Sexual hormone binding globulin | Multiple time points up to treatment day 84
Number of patients with adverse events | Up to 84 days
Number of patients with abnormal safety laboratory | Up to 84 days
Time course of follicle-stimulating hormone | Day 27 of pretreatment cycle to treatment day 83
  Serum concentration of follicle-stimulating hormone (FSH)
Time course of luteinizing hormone | Day 27 of pretreatment cycle to treatment day 83
  Serum concentration of luteinizing hormone (LH)

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (7):
- Russia (5):
  - Irkutsk
  - Krasnodar
  - Moscow
  - Saint Petersburg
  - Smolensk
- Ukraine (2):
  - Kiev
  - Zaporizhzhya